CLINICAL TRIAL: NCT06055829
Title: The Adjustment of Doses in Diabetes Mellitus Can Lead to Fluctuation of Glucose Level in Type I
Brief Title: The Adjustment of Doses in Diabetes Mellitus Type I
Status: Completed | Type: Observational
Sponsor: Liwa College (Other)
Responsible Party: Principal Investigator, Hisham Ibrahim, Dr., Liwa College
Other Study IDs: 4a-V8
Record Dates: First submitted 2023-09-20; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes mellitus, Insulin injection, Patients training
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — Insulin; Blood Glucose

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Drug: Insulin injection and blood glucose — The FreeStyle Libre sensor continuously measures glucose every minute and saves the glucose data. Scan the sensor at least every 8 hours for a full glycemic profile. The below data is displayed after a typical 1-second scan of the FreeStyle LibreLink app or FreeStyle Libre reader via the sensor:
  Other Names: FreeStyle Libre sensor

SUMMARY:
The study was carried out in a diabetic patient who was starting a new approach for treatment. Previously the patient was treated with Novo-mix insulin injection twice per day, the physician decided to change the treatment strategy to be with three doses of novo-rapid insulin injections per day plus one injection of Lantus SoloStar in dinner. For two weeks we were monitoring the blood glucose level by the FreeStyle Libre sensor. Moreover, the right statistical technique was used for data analysis.

DETAILED DESCRIPTION:
In this study a diabetic patient is starting a new approach to treatment. Previously, the patient received Novo-Mix insulin injection twice per day (48 Units in breakfast & 28 Units in dinner). Moreover, the physician decided to change the treatment strategy to be with Novo-Rapid insulin injection three times per day (36 Units in breakfast, 36 Units in lunch & 50 Units in dinner) plus one time injection of Lantus SoloStar (50 Units) in dinner. Thus, for monitoring blood glucose level, we are using the FreeStyle Libre-Link. Moreover. Moreover, FreeStyle Libre sensor continuously measures glucose every time when scanned by the mobile and saves the glucose data in the library. Moreover, scanning the FreeStyle Libre sensor with a phone or the reader measures the glucose levels from the interstitial fluid, a thin layer of fluid that surrounds the cells of the tissues in the skin of the patient [4]. The Scan was done every 1-2 hours for a full glycemic profile.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patient

Exclusion Criteria:

* Normal patient

Ages: 41 Years to 41 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study was carried out in a diabetic patient who was starting a new approach for treatment. Previously the patient was treated with Novo-mix insulin injection twice per day, the physician decided to change the treatment strategy to be with three doses of novo-rapid insulin injections per day plus one injection of Lantus SoloStar at dinner.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2022-10-24 (Actual); Primary Completion 2022-11-06 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
Glucose level | Two weeks
  the physician decided to change the treatment strategy to be with Novo-Rapid insulin injection three times per day (36 Units in breakfast, 36 Units in lunch & 50 Units in dinner) plus one injection of Lantus SoloStar (50 Units) at dinner.

CONTACTS AND LOCATIONS:
Locations (1):
- Hisham Ibrahim, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Yes
The results
Supporting Information: CSR
Time Frame: Open
Access Criteria: any one
URL: https://drive.google.com/drive/u/0/folders/1fy34R987DpzBqomlzb84JqUzUvyELXRu

REFERENCES:
- [Background] Shi XY, Zhang K, Zhang L. [Type 1 diabetes millitus following short-term recombinant interferon therapy in patient with chronic hepatitis C]. Zhonghua Nei Ke Za Zhi. 2018 Jul 1;57(7):524-525. doi: 10.3760/cma.j.issn.0578-1426.2018.07.012. No abstract available. Chinese. PMID 29996274
- [Background] Nauck MA, Quast DR, Wefers J, Meier JJ. GLP-1 receptor agonists in the treatment of type 2 diabetes - state-of-the-art. Mol Metab. 2021 Apr;46:101102. doi: 10.1016/j.molmet.2020.101102. Epub 2020 Oct 14. PMID 33068776
- See also: FreeStyle Libre information — http://www.freestyle.abbott/ae-en/home.html
- See also: NovoRapid information — https://www.ema.europa.eu/en/documents/overview/novorapid-epar-summary-public_en.pdf